CLINICAL TRIAL: NCT03384199
Title: The Impact of Dose Escalation Using Gold Markers in Image Guided Volumetric Modulated Arc Radiotherapy to the Focal Lesion Micro Boost of Localized Prostate Cancer
Brief Title: Dose Escalation Using Fiducial Markers in Image Guided Volumetric Modulated Arc Therapy to the Focal Lesion Micro Boost of Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Radwa Fawzy, assistant Lecturer of Clinical Oncology, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Prostate
Record Dates: First submitted 2016-08-21; First posted 2017-12-27 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Prostatic Adenocarcinoma
Keywords: Localized Prostate; VMAT; Dose escalation; Fiducial marker; Focal Lesion; Random error during dose escalation radiotherapy; fiducial marker image guided technique

STUDY DESIGN:
Intervention Model Description: VMAT dose escalation protocol with image guided fiducial markers
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escaltion (Experimental): insertion of 3 fiducial markers, prostate will receive 78 Gy with dose escalation to prostate focal lesion up to 87 Gy
  Interventions: Radiation: Dose escalation to prostate focal lesion

INTERVENTIONS:
Radiation: Dose escalation to prostate focal lesion — For each patient the radio-opaque marker (used for treatment verification) will be inserted by ultrasound guidance & local anaesthetic with an 17ga x 30cm brachytherapy needle that has 1.2mm x 3mm one gold marker. The ultrasound probe (as used for transrectal biopsy) will be introduced rectally with the patient in the left lateral position. After measuring the volume of the prostate and determining the desired position (preferably in the corpus of prostate), three gold markers will be inserted as follows: one into right side, one into left side of the base and the third in the apex of the prostate

SUMMARY:
Gold markers implanted in the prostate are used frequently for position verification of the prostate during external-beam radiotherapy. By using the markers as a surrogate for the prostate itself, not only set-up errors, but also the internal motion of the prostate relative to the bony anatomy can be identified.

It is thus believed that escalated dose marker guided radiotherapy should result in better biochemical control compared to conventional external beam radiotherapy, with a similar or lower incidence of toxicity. However, clinical data to support this is still limited. The purpose of this study is to directly compare late toxicity as well as biochemical control between patients treated with dose escalated marker guided radiotherapy versus conventional dose non-marker guided radiotherapy who has otherwise been treated with similar radiotherapy planning techniques and equipment.

Prostate magnetic resonance imaging has undergone several technical improvements and shows promises for prostate tumor detection and localization. In addition to morphological information, magnetic resonance imaging allows an estimation of physiological properties of tissues. Diffusion-weighted magnetic resonance imaging is sensitive to restriction of diffusion of water molecules, and dynamic contrast enhanced magnetic resonance imaging can analyze tissue micro vascular properties. Multi para metric magnetic resonance imaging combining Diffusion-weighted and Dynamic contrast enhanced has demonstrated its value in distinguishing malignant from benign prostate tissue.

Higher radiation dose levels were consistently associated with improved biochemical control outcomes and reduction in distant metastases. Radiation dose was one of the important predictors of long-term biochemical tumor control. Dose levels < 70.2 Grey and 70.2-79.2 Grey were associated with 2.3 and 1.3-fold increased risks of pro static specific antigen relapse compared with higher doses. However, further dose escalation to the whole gland is limited due to an unacceptable high risk of acute and late toxicity. Moreover, local recurrences often originate at the location of the macroscopic tumor, so boosting the radiation dose at the macroscopic tumor within the prostate might increase local control. A reduction of distant metastases and improved survival can be expected by reducing local failure. Treating the dominant focus or boosting the dose to this area while reducing the dose to as much healthy tissue as possible has significant potential for improving treatment.

DETAILED DESCRIPTION:
Thirty consecuative loclized prostate cancer patients will be recruited according to inclusion & exclusion criteria. Once the patient meets the selection criteria stratification will be done according to the following risk group classification:

Stage Gleason score PSA Low risk T1-T2a 2-6 < 10 ng/mL Intermediate risk T2b-T2c 7 10-20 ng/mL High risk T3a 8-10 > 20 ng/mL

The patient will receive 2-6 months of neo adjuvant hormonal treatment, followed with concomitant hormonal treatment during the radiation course for intermediate and high risk groups then adjuvant hormonal for 2-3 years in the high risk group.

For each patient the radio-opaque marker (used for treatment verification) will be inserted by ultrasound guidance & local anesthetic with an 17 GA x 30 cm brachy therapy needle that has 1.2 mm x 3 mm one gold marker. The ultrasound probe (as used for trans rectal biopsy) will be introduced rectally with the patient in the left lateral position. After measuring the volume of the prostate and determining the desired position (preferably in the corpus of prostate), three gold markers will be inserted as follows: one into right side, one into left side of the base and the third in the apex of the prostate. All patients will receive a course of preventive antibiotic treatment that consists of ciprofloxacine 500 mg BID, 1 day before implantation and 4 consecutive days. Patients under anti-platelet therapy will be told to stop the medication 5 days before implantation.

CT images will be done within 5 days of markers insertion in the same treatment supine position with Knee & ankle support. CT images will be taken in 1.25 mm slice thickness from the top of the 4th lumbar vertebrae to ischial tuberosities. Patients will be asked to evacuate bowels prior to scanning, and bladder will be kept comfortably full by drinking two glasses of water (250-500 ml) 30 min prior to the scan.

The reference marks, one mid line and two lateral, will be placed at the level of the upper border of the symphysis pubis or iliac crest. No contrast will be used so as to avoid the dose artifact by it during treatment planning and dose calculation.

Multi parametric magnetic resonance imaging combing Diffusion-weighted & Dynamic contrast enhanced with intravenous contrast will be done prior to Marker insertion with the sequence of: axial T1 & T2, coronal T2 & spare, post contrast dynamic axial & sagittal and diffusion with ADC. The views of MRI images will be in 1.25 mm thickness with 0 gap. Fusion of both CT images & MRI images will be done using manual registration guided by bony landmarks.

Delineation of clinical target volumes & risk organs will be done on CT images guided with MRI fused images according to Radiation therapy oncology group criteria. MRI T2 weighted images will guide the pro static delineation from base to apex, with more accurate identification of the apex compared to CT. Also Diffusion-weighted with Dynamic contrast enhanced magnetic resonant imaging will be of value for identification of dominant focal lesion of the prostate.

The patient will be treated with radical radiotherapy to prostate 78 Gray/35# (2.2 Gray/#) with simultaneous integrated boost to focal lesion 87.5 Grey/35# (2.5 Gray/#). Lymph node 60 Grey if positively involved. Seminal vesicle will receive 78 Gray if involved & 54 Gray if not. Roche formula will be used to estimate lymph node & seminal vesicle involvement if more than 15%:

* Seminal vesicle involvement (%) = PSA + [10× (Gleason-6)]
* Pelvic lymph node involvement = 2/3 × PSA + [10× (Gleason score -6)]

Constrains for organs at risk will be followed according to QUANTEC. Plan acceptance for Planning target volume of the targets will be done as follows:

* D 95(95% of the prescribed dose) must be received by at least 95% of the planning target volume.
* D max (dose received by 2% of the volume) should not exceed 107% and should be inside the clinical target volume.
* D min (dose received by 98% of the volume) should not be less than 90% and should be outside the clinical target volume.

In addition to the standard quality assurance procedures carried out for any radiation technique, such as dose output calibration, ISO-center and Multi-leaf collimator verification, V MAT patients will undergo specific pretreatment quality assurance measures to check ISO-center absolute dose (using ionization chamber and slap phantom) and dose (using portal image and portal dosimeter module on the planning system).

Position verification will be done guided with implanted gold markers with daily portal imaging (AP & lateral) correction protocol in mediolateral, superior-inferior & inward-outward directions. The portal correction images will be verified daily to detect average shifts in the three directions using 2D-2D match & Marker Match. Random or inter-fraction errors which are deviations between different fractions will be taken weekly during a treatment series. Systematic errors Which are deviations between the planned patient position and the average patient position of a course of fractional therapy will be taken in the first three settings. The mean and standard deviation (SD) of the systematic error and SD of random errors will be analyzed. To represent true magnitude of errors, the absolute value of the deviations will be also considered. These means will be used in calculations of the off-line treated Dose-Volume Histogram versus Planned Dose-Volume Histogram and in measurement of systemic & random error to define reasonable planning target volume.

Follow up of the patients will be done with mean of 12 months to detect biochemical control & disease free survival. PSA & pelvic ultrasound will be done every 3 months for first 2 years then every 6 months for 3-5 years. Genito-urinary, gastro-intestinal & hematological toxicity will be assessed using Radiation Therapy Oncology Group toxicity score & patient reported out coming will be assessed using questionnaire (validated Arabic translation) every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Performance status ECOG: 0-2
2. Pathologically proven prostatic adenocarcinoma.
3. Localized prostate cancer (Gleason's score: 2-10, Baseline serum prostatic antigen: >4 ng/dl, T1a-T3b).
4. No extra prostatic invading adjacent structures.
5. Adequate hematological, renal & hepatic profile.
6. Insertion of more than one fiducial marker in the prostate.
7. Patient did verbal & written consent and adherence to treatment.

Exclusion Criteria:

1. Patient weight >130 kg.
2. Performance status EGOG: 3-4.
3. Distant metastasis.
4. Previous pelvic radiotherapy.
5. Previous prostatectomy.
6. Urinary bladder stones.
7. General contraindications for MRI (i.e. cardiac pacemaker, metal implants or history of severe allergic reaction after administration of contrast agent).
8. Concomitant neoplastic disease or previous anti neoplastic therapy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Measurement of systemic error in mm and random error in cm in the different three direction X-Y-Z | 12 months
  Position verification will be done guided with implanted gold markers with daily portal imaging (AP & lateral) correction protocol in mediolateral, superior-inferior & inward-outward directions by mm for 35 fraction. The off-line portal pre-correction images will be verified daily to detect average shifts in the three diresctions. Random or inter-fraction errors which are deviations between different fractions will be taken weekly during a treatment series. Systematic errors Which are deviations between the planned patient position and the average patient position of a course of fractioned therapy will be taken in the first three settings. The mean and standard deviation (SD) of the systematic error and SD of random errors will be analyzed.

SECONDARY OUTCOMES:
Biochemical relapse of PSA above normal level 4 ng/dl | 12 months
  Follow up of the patients will be done every 3 months up to 12 months to detect biochemical control by PSA measuring. PSA & pelvic ultrasound.
subjective toxicity assessment | 12 months
  Genito-urinary & gastro-intestinal will be assessed using RTOG toxicity score weekly during radiotherapy sessions.
Objective toxicity assessment | 12 months
  Patient reported out coming will be assessed using FACIT questionnaire (validated Arabic translation) every 3 months up to 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Radwa Fawzy Saleh Ahmed, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Abstract and paper publication